CLINICAL TRIAL: NCT03829150
Title: Anti-Helicobacter Pylori Therapy With Dexlansoprazole MR-Based Concomitant Quadruple Therapy- A Prospective Randomized Trial
Brief Title: Dexlansoprazole MR-Based Concomitant Quadruple Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Seng-Kee Chuah, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG8F1421
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: non-bismuth containing quadruple therapy
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexlansoprazole MR group (Experimental): Dexlansoprazole MR 60 mg qd.,clarithromycin 500 mg bid., amoxicillin 1 g bid. and metronidazole 500 mg bid. for 7 days
  Interventions: Drug: Dexlan; Drug: Amoxicillin; Drug: Clarithromycin 500mg; Drug: Metronidazole
- lansoprazole group (Experimental): Lansoprazole 30 mg bid., clarithromycin 500 mg bid., amoxicillin 1 g bid. and metronidazole 500 mg bid. for 7 days
  Interventions: Drug: Dexlan; Drug: Amoxicillin; Drug: Clarithromycin 500mg; Drug: Metronidazole

INTERVENTIONS:
Drug: Dexlan — Dexlansoprazole MR 60 mg qd for 7 days
  Other Names: Dexlansoprazole MR
Drug: Amoxicillin — Amoxicillin (Amolin) 1 g bid. for 7 days
  Other Names: Amolin
Drug: Clarithromycin 500mg — clarithromycin (Klaricid) 500 mg bid for 7 days
  Other Names: Klaricid
Drug: Metronidazole — Metronidazole (Flagyl) 500 mg bid daily for 7 days
  Other Names: Flagyl

SUMMARY:
Background:

Recommended proton pump inhibitor (PPI)-clarithromycin-amoxicillin or metronidazole treatment for 7 to14 days is the first choice treatment for H pylori infection. The eradication rate of the standard triple therapy has generally declined to unacceptable levels (i.e., 80% or less) recently because the increasing incidence of clarithromycin-resistant strains of H. pylori. Standard triple therapies should be abandoned in the areas with clarithromycin resistance ≥ 20%. The investigators have proven that 7-day Concomitant therapy can achieve a promising success rate of >90 % in the presence of clarithromycin resistance. However, high dose PPI is needed with a dosage of twice daily but when a dual delayed release formulation PPI in capsules for oral administration (Dexlansoprazole MR), a once daily dose may be needed only. The capsules contain dexlansoprazole in a mixture of two types of enteric-coated granules with different pH-dependent dissolution profiles. It suppresses gastric acid secretion via inhibition of the proton pump in the gastric parietal cell, which blocks the final step of acid production. Thus, it improves acid suppression and offer benefits over conventional single release PPI formulations. by prolonging optimal plasma concentration and create a favorable condition H. pylori eradication

Aim:

The efficacy of Dexlansoprazole MR-based concomitant quadruple therapy

DETAILED DESCRIPTION:
Background:

Recommended proton pump inhibitor (PPI)-clarithromycin-amoxicillin or metronidazole treatment for 7 to14 days is the first choice treatment for H pylori infection. The eradication rate of the standard triple therapy has generally declined to unacceptable levels (i.e., 80% or less) recently because the increasing incidence of clarithromycin-resistant strains of H. pylori. Standard triple therapies should be abandoned in the areas with clarithromycin resistance ≥ 20%. The investigators have proven that 7-day Concomitant therapy can achieve a promising success rate of >90% in the presence of clarithromycin resistance. However, high dose PPI is needed with a dosage of twice daily but when a dual delayed release formulation PPI in capsules for oral administration (Dexlansoprazole MR), a once daily dose may be needed only. The capsules contain dexlansoprazole in a mixture of two types of enteric-coated granules with different pH-dependent dissolution profiles. It suppresses gastric acid secretion via inhibition of the proton pump in the gastric parietal cell, which blocks the final step of acid production. Thus, it improves acid suppression and offer benefits over conventional single release PPI formulations. by prolonging optimal plasma concentration and create a favorable condition H. pylori eradication

Aim:

The efficacy of Dexlansoprazole MR-based concomitant quadruple therapy

Methods:

Two hundred and two consecutive H. pylori-infected participants are randomly assigned to a 7-day Dexlansoprazole MR-based non-bismuth quadruple therapy (Dexlansoprazole MR 60 mg qd.,clarithromycin 500 mg bid., amoxicillin 1 g bid. and metronidazole 500 mg bid. for 7 days) or a 7-day lansoprazole-based non-bismuth quadruple therapy (Lansoprazole 30 mg bid. , clarithromycin 500 mg bid., amoxicillin 1 g bid. and metronidazole 500 mg bid. for 7 days). Participants are asked to return at the 2nd week to assess drug compliance and adverse events. Repeated endoscopy with rapid urease test, histological examination is performed at the 8th week after the end of anti- H. pylori therapy. If participants refuse follow-up endoscopy, urea breath tests are conducted to assess H. pylori status. The rates of eradication are analyzed by intention-to-treat and per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

H. pylori-infected outpatients with endoscopically proven peptic ulcer diseases or gastritis.

Exclusion Criteria:

1. Previous H. pylori-eradication therapy
2. ingestion of antibiotics, bismuth, or PPIs within the prior 4 weeks
3. patients with allergic history to the medications used
4. patients with previous gastric surgery
5. the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
6. pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
The rates of H.pylori eradication | 8 weeks
  The primary outcome variables were the rates of eradication. Chi-square test with or without Yates correction for continuity and Fisher's exact test were used when appropriate to compare the major outcomes between groups. A P value less than 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Seng-Kee Chuah, MD, Principal Investigator — Kaohsiung Chang Gung Memorial Hospital,Taiwan
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital,Taiwan, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Tai WC, Liang CM, Bi KW, Kuo CM, Lu LS, Wu CK, Yang SC, Kuo YH, Lee CH, Huang CF, Hsu CN, Hsu PI, Wu DC, Hu TH, Wu KL, Chuah SK. A comparison between dexlansoprazole modified release-based and lansoprazole-based nonbismuth quadruple (concomitant) therapy for first-line Helicobacter pylori eradication: a prospective randomized trial. Infect Drug Resist. 2019 Sep 16;12:2923-2931. doi: 10.2147/IDR.S213998. eCollection 2019. PMID 31571945